CLINICAL TRIAL: NCT05133336
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Phase 2b/3 Study to Evaluate the Efficacy and Safety of Saroglitazar Magnesium in Subjects With Primary Biliary Cholangitis
Brief Title: Saroglitazar Magnesium for Treatment of Primary Biliary Cholangitis
Acronym: EPICS-III
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.21.001
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Primary Biliary Cholangitis
Keywords: Saroglitazar Magnesium; Primary Biliary Cholangitis; PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — saroglitazar

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-blind, Placebo controlled, Phase 2b/3 Safety and Efficacy Study . Initially, 192 subjects (64 subjects in each treatment arm) were planned be randomised in a ratio of 1:1:1 in Saroglitazar Magnesium 1 mg, Saroglitazar Magnesium 2 mg, and Placebo arm, respectively. After an optimal dose selection, the subjects are randomised in 2:1 ratio of Saroglitazar Magnesium 1 mg or placebo. There would be approximately 140 evaluable subjects (90 of Saroglitazar 1 mg and 50 of placebo arm)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saroglitazar Magnesium 2 mg (Experimental): Subjects who received Saroglitazar Magnesium 2 mg tablet orally administered once daily in the morning before breakfast are switched to Saroglitazar Magnesium 1 mg for remaining of the treatment period
  Interventions: Drug: Saroglitazar Magnesium 1 mg; Drug: Saroglitazar Magnesium 2 mg
- Saroglitazar Magnesium 1 mg (Experimental): Saroglitazar Magnesium 1 mg tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment (52 weeks).
  Interventions: Drug: Saroglitazar Magnesium 1 mg
- Placebo (Placebo Comparator): Placebo tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment (52 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar Magnesium 1 mg — Subjects randomized to Saroglitazar Magnesium 1 mg arm will receive Saroglitazar Magnesium 1 mg treatment for the entire treatment period up to Week 52.
  Arms: Saroglitazar Magnesium 1 mg; Saroglitazar Magnesium 2 mg
Drug: Saroglitazar Magnesium 2 mg — Subjects randomized to Saroglitazar Magnesium 2 mg arm are switched to Saroglitazar Magnesium 1 mg treatment up to Week 52
  Arms: Saroglitazar Magnesium 2 mg
Drug: Placebo — Subjects randomized to placebo arm will receive placebo treatment for the entire treatment period up to Week 52.
  Arms: Placebo

SUMMARY:
Saroglitazar Magnesium 1 mg and 2 mg tablets for treatment of subjects with Primary Biliary Cholangitis (PBC)

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Placebo controlled, Phase 2b/3 Study to Evaluate the Efficacy and Safety of Saroglitazar Magnesium in Subjects with Primary Biliary Cholangitis

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 75 years of age, both inclusive at screening.
2. Subjects on ursodeoxycholic acid (UDCA) for at least 12 months at a therapeutic dose (at least 13 mg/kg per day) and a stable dose for 6 months prior to Screening Visit and having ALP ≥ 1.67 x ULN.

   OR Subjects who are unable to tolerate UDCA and did not receive UDCA for at least 3 months prior to the date of screening and having ALP ≥ 1.67 x ULN.
3. History of confirmed PBC diagnosis, based on American Association for the Study of Liver Disease [AASLD] and European Association for Study of the Liver [EASL] Practice Guidelines, as demonstrated by the presence of at least ≥ 2 of the following 3 diagnostic factors:

   * History of elevated ALP levels for at least 6 months prior to screening
   * Positive anti-mitochondrial antibodies (AMA) titer OR positive PBC specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex]) if AMA is negative
   * Liver biopsy consistent with PBC
4. ALP ≥ 1.67 x ULN at both Visits 1 and 2 and < 30% variance between the levels from Visit 1 to Visit 2
5. Total bilirubin < 2 x ULN at screening (Visit 1)
6. Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

1. Consumption of 2 standard alcohol drinks per day if male and 1 standard alcohol drink per day if female for at least 3 consecutive months (12 consecutive weeks) within 5 year before screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor).
2. History or presence of other concomitant liver diseases at screening:

   1. Chronic hepatitis B or C virus (HBV, HCV) infection. (Note: However, If the subject has been treated for the HCV infection and has been cured for a duration of more than 2 years from screening, such subjects can be enrolled in the study)
   2. Primary sclerosing cholangitis (PSC).
   3. Alcoholic liver disease.
   4. Autoimmune hepatitis (AIH) indicative of PBC with overlap syndrome.

Note: The Paris criteria are commonly used to define the presence of PBC with features of AIH and have been endorsed by EASL and AASLD. According to these criteria, a diagnosis can be made in a patient with PBC as follows:

At least two of the following:

I. ALP > 2 x ULN or GGT > 5 x ULN. II. AMA positive III. Florid bile duct lesion on histology. AND

At least two of the following three features:

I. ALT > 5 x ULN. II. Immunoglobulin G serum levels > 2 x ULN or smooth muscle autoantibody positive.

III. Moderate to severe interface hepatitis on histology. e. Hemochromatosis. f. Non-alcoholic steatohepatitis (NASH) on historical biopsy. 3.Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, ascites requiring treatment, encephalopathy, known large esophageal varices or history of variceal bleeding within one year prior to screening or history of hepatorenal syndrome.

5.Medical conditions that may cause non-hepatic increases in ALP (e.g., Paget's disease) or which may diminish life expectancy to < 2 years, including known cancers.

6.Use of thiazolidinediones or fibrates (within 12 weeks prior to screening). 7.Use of obeticholic acid (OCA), azathioprine, cyclosporine, methotrexate, mycophenolate, pentoxifylline, budesonide and other systemic corticosteroids (Note: Prednisone dose should not be more than 10 mg per day); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid, or nitrofurantoin) (within 12 weeks prior to screening).

9.History of bowel surgery (gastrointestinal [bariatric] surgery in the preceding 1 year or undergoing evaluation for gastrointestinal surgery (bariatric surgery for obesity, extensive small-bowel resection) or orthotopic liver transplant (OLT) or listed for OLT.

10.Type 1 diabetes mellitus. 11.Unstable cardiovascular disease, including:

a. Unstable angina, (i.e., new or worsening symptoms of coronary heart disease in the 12 weeks before screening and throughout the Screening Period), acute coronary syndrome in the 24 weeks before screening and throughout the Screening Period, acute myocardial infarction in the 12 weeks before screening and throughout the Screening Period or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, in the 24 weeks before screening and throughout the Screening Period.

b. History/current unstable cardiac dysrhythmias. c. Uncontrolled hypertension at screening. d. Stroke or transient ischemic attack in the 24 weeks before screening. 12.History of intracranial hemorrhage, arteriovenous malformation, bleeding disorder, coagulation disorders, or screening blood tests that, in the opinion of the Investigator, indicate altered coagulability (e.g., PT, INR, aPTT) at screening.

13.An uncontrolled thyroid disorder

1. Uncontrolled hyperthyroidism: defined as any history of hyperthyroidism that has either not been treated with either radioactive iodine and/or surgery or that has been treated with radioactive iodine and/or surgery, but has required ongoing continuous or intermittent use of thyroid hormone synthesis inhibitors (i.e., methimazole or propylthiouracil) in the 24 weeks before screening.
2. Uncontrolled hypothyroidism: defined as initiation of thyroid hormone replacement therapy or dose adjustment of replacement therapy in the 12 weeks before screening.

   14.History of myopathies or evidence of active muscle disease demonstrated by CPK ≥ 5 x ULN at screening.

   15.Subjects whose ALT, AST, or ALP exceeds by more than 50% on Visit 2 reading compared to Visit 1. Note: If the ALT, AST, or ALP values on Visit 2 exceed by more than 50% from Visit 1, then a third value will be measured (within 1- 2 weeks) to assess for the trend. If the third value shows continued increase ≥ 10%, then subject is considered ineligible for randomization.

   16.Any of the following laboratory values at screening:

a. Platelets < 50 × 109/L b. Albumin < 2.8 g/dL c. eGFR < 45 mL/min/1.73 m2 d. ALP > 10 x ULN e. ALT or AST > 250 U/L 17.Participation in another interventional clinical study and receipt of any other investigational medication (within 12 weeks prior to randomization up to end of study).

18.History of malignancy in the past 5 years and/or active neoplasm with the exception of resolved superficial non-melanoma skin cancer.

19.Contraindications to Saroglitazar Magnesium or has any conditions affecting the ability to evaluate the effects of Saroglitazar Magnesium.

20.Known allergy, sensitivity, or intolerance to the study drug, comparator, or formulation ingredients.

21.Pregnancy-related exclusions, including:

a. Pregnant/lactating female (including positive pregnancy test at screening). b. Pregnancy should be avoided by male and female subjects either by true abstinence or the use of an acceptable effective contraceptive measures for the duration of the study and for at least 1 month after the end of the study treatment. Refer Appendix 8 Contraceptive Guidance 22.History or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the Investigator, unsuitable for the study (such as poorly controlled psychiatric disease, HIV, coronary artery disease, or active gastrointestinal conditions that might interfere with drug absorption).

23.Cirrhosis with Child-Pugh-Turcotte (CPT) Class B or C having score of 7 or above at screening 24.Subjects with Model for End Stage Liver Disease (MELD 3.0) score of 12 or above

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with biochemical response based on the composite endpoints of ALP and total bilirubin | From baseline to week 52
  ALP < 1.67 x ULN, ≥ 15% decrease in ALP relative to baseline, and total bilirubin ≤ ULN or direct bilirubin ≤ ULN in subjects with known Gilbert's syndrome

SECONDARY OUTCOMES:
Proportion of subjects with complete normalization of ALP. | From baseline to week 52
  ALP≤ULN
Pruritis assessed by 5 D itch scales | From baseline to Week 24 and Week 52
  Change from baseline in 5-D itch score
Proportion of subjects with biochemical response based on the composite endpoints of ALP and total bilirubin | From baseline to Weeks 4, 8, 16, and 24.
  ALP < 1.67 x ULN, ≥ 15% decrease in ALP, and total bilirubin ≤ ULN or direct bilirubin ≤ ULN in subjects with known Gilbert's syndrome
Proportion of subjects change from baseline in ALP | From baseline to Weeks 24 and 52.
  ALP improvement of at least 15%, 30%, 40%, and 50% Absolute and percent change from baseline in ALP values
Quality of life assessed by the PBC 40 questionnaire | From baseline to Weeks 16, 24, and 52.
  Change from baseline in quality of life (PBC 40) questionnaire domains (total score and domain score)
Improvement in liver stiffness measurement (LSM) of at least 25% relative to baseline assessed by Liver elastography/FibroScan® | From baseline to Weeks 24 and Week 52
  Proportion of subjects with a decrease in LSM of at least 25%
To effect on liver enzymes | From baseline at Weeks 16, 24, and 52.
  Change from baseline in liver enzyme parameters (ALT, AST, GGT, and total bilirubin [direct and indirect bilirubin])
The effect on liver enzymes | From baseline to week 24 and week 52
  Change from baseline in serum bile acids
The effect on lipid parameters | From baseline to weeks 24 and 52
  Change from baseline in lipid parameters (TG, LDL-C, HDL-C, VLDL-C, total cholesterol, and non-HDL-C)

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, MD, Study Director — Zydus Therapeutics Inc.
Locations (57):
- United States (31):
  - Zydus US007, Birmingham, Alabama
  - Zydus US021, Tucson, Arizona
  - Zydus US013, Los Angeles, California
  - Zydus US011, Pasadena, California
  - Zydus US043, Sacramento, California
  - Zydus US022, Aurora, Colorado
  - Zydus US037, New Haven, Connecticut
  - Zydus US027, Jacksonville, Florida
  - Zydus US006, Lakewood Rch, Florida
  - Zydus US005, Miami, Florida
  - Zydus US028, Sarasota, Florida
  - Zydus US019, Tampa, Florida
  - Zydus US020, Marietta, Georgia
  - Zydus US001, Indianapolis, Indiana
  - Zydus US034, Iowa City, Iowa
  - Zydus US036, Marrero, Louisiana
  - Zydus US023, Rochester, Minnesota
  - Zydus US030, St Louis, Missouri
  - Zydus US024, Omaha, Nebraska
  - Zydus US038, Manhasset, New York
  - Zydus US035, Rochester, New York
  - Zydus US002, Charlotte, North Carolina
  - Zydus US014, Cincinnati, Ohio
  - Zydus US015, Philadelphia, Pennsylvania
  - Zydus US004, Houston, Texas
  - Zydus US042, Houston, Texas
  - Zydus US031, Murray, Utah
  - Zydus US016, Charlottesville, Virginia
  - Zydus US041, Newport News, Virginia
  - Zydus US039, Richmond, Virginia
  - Zydus US033, Seattle, Washington
- Argentina (10):
  - Zydus AR004, Buenos Aires
  - Zydus AR009, Buenos Aires
  - Zydus AR001, Buenos Aires
  - Zydus AR005, Buenos Aires
  - Zydus AR013, Buenos Aires
  - Zydus AR007, Buenos Aires
  - Zydus AR006, Buenos Aires
  - Zydus AR012, Buenos Aires
  - Zydus AR003, Buenos Aires
  - Zydus AR010, Santa Fe
- Zydus IS001, Reykjavik, Iceland
- Turkey (Türkiye) (15):
  - Zydus TR014, Adana
  - Zydus TR016, Altındağ
  - Zydus TR004, Ankara
  - Zydus TR005, Bursa
  - Zydus TR017, Cebeli
  - Zydus TR008, Gaziantep
  - Zydus TR009, Istanbul
  - Zydus TR010, Istanbul
  - Zydus TR003, Istanbul
  - Zydus TR001, Istanbul
  - Zydus TR002, Izmir
  - Zydus TR013, Izmir
  - Zydus TR011, Kocaeli
  - Zydus TR015, Melikgazi
  - Zydus TR006, Mersin